CLINICAL TRIAL: NCT00989105
Title: A Cancer Research UK Phase I Trial of 99mTc Demobesin-4 (a Diagnostic Radiopharmaceutical) Given Once Via Bolus Intravenous Injection for Imaging of Prostate Cancer
Brief Title: Technetium Tc 99m Demobesin-4 for Imaging Procedures in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000650867; UKM-ICRF-CR0402-11; CRUK-CR0402-11; EUDRACT-2007-005324-32; EU-20981
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Immunohistochemistry; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: computed tomography
Procedure: magnetic resonance imaging
Procedure: single photon emission computed tomography
Radiation: technetium Tc 99m demobesin-4

SUMMARY:
RATIONALE: Diagnostic procedures, such as technetium Tc 99m demobesin-4 followed by single-photon emission computer tomography, CT scan, and MRI, may help find prostate cancer and learn the extent of disease.

PURPOSE: This phase I trial is studying the side effects of technetium Tc 99m demobesin-4 and to see how well it works for imaging procedures in patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety of technetium Tc 99m (^99mTc) demobesin-4 (DB4) in patients with prostate cancer.
* To assess the biodistribution of ^99mTc DB4 in these patients.
* To assess the pharmacokinetics of ^99mTc DB4 in these patients.

Secondary

* To assess the performance of ^99mTc DB4 in detecting metastatic spread of prostate cancer in these patients.

Tertiary

* To compare uptake of ^99mTc DB4 with levels of expression in gastrin-releasing peptide receptor in prostate tumor samples and lymph node specimens.

OUTLINE: Patients are stratified according to diagnosis (cancer confined to prostate vs locally advanced disease vs metastatic disease).

Patients receive technetium Tc 99m (^99mTc) demobesin-4 (DB4) IV bolus over 1 minute and undergo imaging by single photon emission computer tomography, CT scan, and/or MRI up to 3 hours after infusion. Some patients undergo radical prostatectomy or surgical pelvic lymph node biopsies.

Blood and urine samples are collected at 5, 10, 20, 30, and 45 minutes at baseline and at 1, 2, 3, 4, and 6 hours after ^99mTc DB4 IV infusion for pharmacokinetic studies. Tumor tissue samples obtained during radical prostatectomy and surgical lymph node biopsies are analyzed for gastrin-releasing peptide receptor by IHC.

After completion of study intervention, patients are followed for up to 28 days.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer meeting 1 of the following criteria:

  * Disease confined to the prostate that is to be treated with radical prostatectomy after imaging
  * Locally advanced disease that is to be treated with radiotherapy

    * Patients must agree to undergo surgical pelvic lymph node staging to assist with determination of radiation fields
  * Metastatic disease at initial diagnosis or recurrent or progressive disease

    * Patients receive standard of care

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Neutrophils ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 times ULN
* Must be registered with the Cancer Research UK Drug Development Office
* Capable of cooperating with imaging procedure and follow-up
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* Not at high medical risk because of non-malignant systemic disease, including active uncontrolled infection
* No history of recent significant cardiac arrhythmia
* No prior NYHA class III-IV cardiac disease or concurrent congestive heart failure
* No other condition that, in the Investigator's opinion, would not make the patient a good candidate for the clinical trial

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No chemotherapy or radiotherapy prior to or within 2 weeks of study therapy
* No prior major thoracic and/or abdominal surgery from which the patient has not yet recovered
* No other concurrent investigational drugs
* Concurrent anticancer therapy allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Causality of each adverse events as assessed by NCI CTCAE v. 3.0
Biodistribution of radioactivity of 99mTc DB4 by gamma-camera imaging
Pharmacokinetics of 99mTc DB4 in blood and urine and assessment of decline over 6 hours

SECONDARY OUTCOMES:
Performance of 99mTc DB4 gamma-camera imaging compared with conventional imaging (CT scan and/or MRI)
Levels of expression in gastrin-releasing peptide in prostate tumor samples and lymph node specimens

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Avril, MD, Principal Investigator — St. Bartholomew's Hospital
Locations (1):
- Saint Bartholomew's Hospital, London, England, United Kingdom